CLINICAL TRIAL: NCT05343572
Title: Bone Marrow Derived Stem Cells Mobilization for Treatment of Asherman's Syndrome, Atrophic Endometrium, and Recurrent Implantation Failure
Brief Title: Bone Marrow Derived Stem Cells Mobilization for Treatment of Abnormal Endometrium
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hugh Taylor (Other)
Responsible Party: Sponsor-Investigator, Hugh Taylor, Chair of Obstetrics, Gynecology and Reproductive Sciences, Yale University
Organization: Yale University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000026217; No NIH funding (Other: 11.15.23)
Record Dates: First submitted 2022-04-11; First posted 2022-04-25 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Asherman Syndrome; Atrophic Endometrium; Recurrent Implantation Failure
Keywords: bone marrow derived stem cells
MeSH Terms: conditions — Gynatresia | interventions — plerixafor

STUDY DESIGN:
Intervention Model Description: This is a pilot, open-label, non-randomized study to investigate the use of autologous bone marrow derived stem cells (peripheral mobilization) for cell-based therapy in treating AS, AE, and RIF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Endometrial Disorders (Experimental): Three groups of patients, with 10 subjects per group:
  1. Asherman's syndrome, as classified by the American Society of Reproductive Medicine (ASRM) by extent of uterine cavity involvement and adhesion type. Specifically, refractory Asherman's syndrome: patients who have had at least one operative hysteroscopy which was unsuccessful.
  2. Atrophic endometrium, as defined by maximal endometrial lining thickness ≤6mm documented in at least 2 cycles on either:
     * Day of luteinizing hormone (LH) surge in natural cycle
     * Day of human chorionic gonadotropin (hCG) trigger in the setting of fresh IVF cycle
     * Day 14 of estradiol in the setting of frozen embryo transfer things (FET) cycles
  3. Recurrent implantation failure, defined as failure to achieve a clinical pregnancy after transfer of at least four good-quality embryos in a minimum of three fresh or frozen transfer cycles in a woman under 40 years
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — A 20mg single dose of PLERIXAFOR is administered subcutaneously the evening prior to scheduled standard of care surgery for women with AS, AE or RIF for peripheral mobilization of stem cells. For subjects weighing >83 kilogram, the dosing is a single dose of 0.24 milligram per kilogram.

SUMMARY:
This study will assess the use of autologous bone marrow stem cells mobilization using 1,1'-[1,4-phenylenebis-(methylene)]-bis-1,4,8,11-tetraazacyclotetradecane (PLERIXAFOR) as an effective medical therapy for the treatment of Asherman's Syndrome (AS), Atrophic Endometrium (AE) and Recurrent Implantation Failure (RIF).

DETAILED DESCRIPTION:
This study will assess the use of autologous bone marrow stem cells mobilization using 1,1'-[1,4-phenylenebis-(methylene)]-bis-1,4,8,11-tetraazacyclotetradecane (PLERIXAFOR) as an effective medical therapy for the treatment of Asherman's Syndrome (AS), Atrophic Endometrium (AE) and Recurrent Implantation Failure (RIF).

Primary Objective:

* To compare endometrial thickness and implantation rates in women with AS, AE, and RIF receiving PLERIXAFOR compared to historic controls that received existing standard of care therapy
* To compare ongoing pregnancy and live birth rates in women with AS, AE, and RIF receiving PLERIXAFOR compared to historic controls that received existing standard of care therapy

Secondary Objectives: (assessed in participants who have not achieved pregnancy as of the timepoint):

- Endometrial thickness prior to treatment with PLERIXAFOR compared to endometrial thickness 3 and 6 months after treatment.

During this study, participants are asked to:

* Refrain from use of non-steroidal anti-inflammatory drugs (NSAIDs) from 2 weeks prior to the start of the surgery/PLERIXAFOR administration, and for the 30 days following surgery/ PLERIXAFOR administration.
* Abstain from intercourse for three months following surgery/PLERIXAFOR administration

  * Assessment of menstrual bleeding pattern before and 3 and 6 months following treatment with PLERIXAFOR
  * Assessment of endometrial blood flow before and 3 and 6 months following treatment with PLERIXAFOR
  * Assessment of endometrial histology three months following treatment with PLERIXAFOR The study intervention consists of administration of PLERIXAFOR the evening prior to scheduled standard of care surgery for women with AS, AE or RIF, for peripheral mobilization of stem cells. PLERIXAFOR is administered via the subcutaneous route, as a single dose of 20mg.

The goal of this study is to determine if the administration of PLERIXAFOR for autologous, peripheral stem cell mobilization and administration will restore endometrial function in women with AS, AE, and RIF, and allow for pregnancy implantation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non pregnant females
* ages ≥18 and ≤40 years old at time of enrollment
* with either AS, AE, or RIF

  1. For AS: surgical history of intrauterine trauma/infection, hypo/amenorrhea, intra-uterine adhesions
  2. for AE: US documentation of persistent, <6mm endometrial thickness
  3. for RIF: failure to achieve a clinical pregnancy after transfer of at least four good-quality embryos in a minimum of three fresh or frozen cycles in a woman under 40 years and currently being treated at Yale Fertility Clinic

Exclusion Criteria:

* Presence of hydrosalpinx (diagnosed by radiographic or ultrasound imaging)
* Endometriosis (diagnosed by previous surgery,)
* Diminished ovarian reserve (AMH<1ng/ml or follicle stimulating hormone (FSH)>10)
* History of genital tuberculosis or any ultrasound evidence of congenital uterine anomaly
* Submucous or intracavitary fibroid, polyps
* Currently pregnant
* Personal history of thrombophilia or sickle cell disease
* Inability to provide informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in endometrial thickness and implantation rates following treatment with Plerixafor at 6 month intervals up to 24 months, compared to controls | Every 6 months from baseline up to 24 months
  Change in endometrial thickness post treatment compared to historic controls that received existing standard of care therapy, measured using ultrasound. Thicker endometrium (>6mm) indicates restoration of endometrial function.

SECONDARY OUTCOMES:
Change in endometrial thickness and implantation rates with Plerixafor in women with AS, AE and RIF at 3 month intervals, compared to baseline/pre-treatment | Every 3 months from baseline up to 24 months
  Change in endometrial thickness and implantation rates with Plerixafor in women with AS, AE and RIF at 3 month intervals, compared to baseline/pre-treatment will be assessed. Less atrophy, less fibrosis, greater blood vessel formation and greater endometrial blood flow on ultrasound, compared to historic controls is indicative of restoration of endometrial function.
Difference in ongoing pregnancy and live birth rates in women with AS, AE and RIF following treatment with Plerixafor at 3 month intervals, compared to baseline/pre-treatment | Every 3 months from baseline up to 24 months
  The difference in ongoing pregnancy and live birth rates in women with AS, AE and RIF following treatment with Plerixafor at 3 month intervals, compared to baseline/pre-treatment will be assessed. Less atrophy, less fibrosis, greater blood vessel formation and greater endometrial blood flow on ultrasound, compared to historic controls is indicative of restoration of endometrial function.
Change in endometrial thickness from baseline after treatment with Plerixafor at month 3 and month 6 for participants that have not achieved pregnancy as of the timepoint | baseline, month 3 and month 6
  Change in endometrial thickness from baseline after treatment with Plerixafor compared to month 3 and month 6 measured using ultrasound. Thicker endometrium (>6mm) indicates restoration of endometrial function.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Taylor, MD, Principal Investigator — Yale University
Locations (1):
- Yale Fertility Center, Orange, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No